CLINICAL TRIAL: NCT03156465
Title: Iowa Cochlear Implant Clinical Research Center Hybrid L24 and Standard Cochlear Implants in Profoundly Deaf Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201109746
Record Dates: First submitted 2017-04-14; First posted 2017-05-17 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Implants, Cochlear; Child; Hearing Loss, Bilateral
MeSH Terms: conditions — Hearing Loss, Bilateral

STUDY DESIGN:
Intervention Model Description: repeated-measure, single-subject experiment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Hybrid L24 and Standard CI (Experimental): Fifteen infants will receive one Nucleus L24 array and a FDA approved standard-length array on contralateral ears.
  Interventions: Device: Hybrid L24

INTERVENTIONS:
Device: Hybrid L24 — Fifteen infants will receive one Nucleus L24 array and a FDA approved standard-length array on contralateral ears.

SUMMARY:
The purpose of this feasibility study is to evaluate whether implantation of one Nucleus L24 electrode array and one FDA approved standard-length device in the contralateral ear can provide useful binaural hearing in pediatric subjects who have bilateral severe to profound hearing loss, meeting the criteria for cochlear implantation. Unlike a conventional cochlear implant, the Nucleus L24 is expected to preserve the regions of the cochlear partition that are apical to the electrode, thus leaving them available for possible future advances in the field of otolaryngology and hearing devices, such as mammalian hair cell regeneration techniques or improved implantable hearing devices. Whether or not this group of children will be able to take advantage of future hair cell regeneration strategies is yet to be determined and will have to wait for future development. At this time there are no accurate imaging strategies available to identify preservation of the scala media. Ultra thin micro CT scanning is in development, however the level of radiation delivery to the subject is too great to be considered for clinical use. When imaging strategies become available to determine cellular structure of the inner ear, they will be applied to this group of subjects. The Nucleus L24 array stimulates the basal turn of the cochlea, in an attempt to preserve the middle and apical regions of the scala media.

DETAILED DESCRIPTION:
The purpose of this feasibility study is to evaluate whether a Nucleus L24 and a FDA approved standard-length device in the contralateral ear can provide useful binaural hearing in pediatric subjects who have bilateral profound hearing loss, meeting the criteria for cochlear implantation. Unlike a conventional cochlear implant, the Nucleus L24 is designed to preserve the regions of the cochlear partition that are apical to the electrode, thus leaving them available for possible future advances in the field of otolaryngology and hearing devices, such as mammalian hair cell regeneration techniques or improved implantable hearing devices. The Nucleus L24 (16 mm) array stimulates the basal turn of the cochlea, in an attempt to preserve the middle and apical regions of the scala media.

The study will be conducted as a repeated-measure, single-subject experiment. A single-subject research design (in which each participant serves as his or her own control) is appropriate because it accommodates the heterogeneity that characterizes hearing-impaired populations. Blinding or masking procedures are not included in the design, as it is not possible to conceal the presence or absence of a cochlear implant from device recipients and/or clinical investigators.

Preoperatively, candidates will be assessed with their current amplification to evaluate their appropriateness for entrance into the study. The candidates' audiometric configuration must meet the above inclusion criteria. That is, the candidate must have a profound sensorineural hearing loss from 250 to 8000 Hz. Prior to testing, the appropriateness of the hearing aid fitting will be assessed and adjustments made if necessary. In cases where amplification has not been used for more than one year, new hearing aids will be fit, worn for a minimum three-month trial and the participants re-evaluated to confirm continuance with the study.

Fifteen infants will receive one Nucleus L24 array and a FDA approved standard-length array on contralateral ears. The investigator will alternate every other subject between the right and left ears as to which ear gets the Nucleus L24. Postoperatively, the right ear only, left ear only, and the bilateral listening modes will be compared with repeated testing through five years of age of the child. These comparisons will help to evaluate the effects of bilateral stimulation using a shorter electrode cochlear implant to possibly preserve the scala media, organ of Corti, and supporting cells for future medical interventions and a standard length implant on the contralateral ear. In addition, the investigator will attempt to compare speech perception and speech/language measure results with age-matched children implanted with standard-length bilateral devices.

ELIGIBILITY:
Inclusion Criteria:

1. Twelve to twenty-four months of age at the time of implantation.
2. Audiometric thresholds for frequencies 250 to 8000 Hz in the profound hearing range bilaterally. The type of hearing loss must be categorized as sensorineural in nature.
3. English spoken as a primary language (mono-lingual English speaking family, where English is the primary language).
4. Willingness to comply with all study requirements.
5. Minimum of three-month hearing aid trial with appropriately fit hearing aids.
6. Patent cochlea and normal cochlear anatomy as shown by a CT scan. It is standard clinical practice to perform a CT scan on any patient pursuing cochlear implantation.

Exclusion Criteria:

1. Medical or psychological conditions that contraindicate undergoing surgery.
2. Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array.
3. Developmental disabilities or other conditions that would prevent or restrict participation in the audiological evaluations and clinical trial.
4. Hearing loss of neural or central origin.
5. Unrealistic expectations on the part of the candidate and/or candidate's family, regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure(s) and prosthetic devices.
6. Unwillingness or inability of the candidate to comply with all investigational requirements.
7. Active middle ear infection.

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2011-09-15 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J Gantz, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hybrid L24 and Standard CI
Started | 11
Completed | 9
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Hybrid L24 and Standard CI
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Infant-Toddler Meaningful Auditory Integration Scale (IT-MAIS)
Description: Parent questionnaire that consists of ten questions regarding a young infant or toddler's auditory behavior, e.g. "Does the child spontaneously respond to his/her name in quiet with auditory cues?" Each question is scored on a five point scale: 0=never, 1=rarely, 2=occasionally, 3=frequently, and 4=always. The aim of this tool is to assess the benefit of the child's personal amplification device(s). This questionnaire is generally used during the cochlear implant work-up to assess hearing aid benefit. It is also used post-cochlear implantation to chart the progress the child is making with his/her cochlear implant when other formalized speech perception tests are not appropriate.
Time Frame: Preoperative through 24 months
Population: some children did not complete the visit
Measure: Mean (Standard Error); unit: percentage out of 40
Arm/Group | Hybrid L24 and Standard CI
Number analyzed (Participants) | 9
percentage out of 40
  Preoperative | 0 (0)
  3 months postoperative: number analyzed (Participants) | 7
  3 months postoperative | 53 (.07)
  6 months postoperative | 64 (.07)
  12 months postoperative: number analyzed (Participants) | 8
  12 months postoperative | 75 (.03)
  24 months postoperative: number analyzed (Participants) | 7
  24 months postoperative | 83 (.05)

2. Primary Outcome: The Early Speech Perception Four Choice Spondee and Monosyllable
Description: Speech perception test that requires the identification of a spondee or monosyllable from a set of four spondees (i.e., French fry, airplane, hotdog, popcorn) or monosyllables (i.e., ball, book, bird, boat), respectively presented in quiet. The CID test will be scored as total number of words correct. It will be administered in both the unilateral and bilateral listening conditions at 70 dB C. This test is given post-operatively until the child scores a ceiling effect which is considered 90% or better in all test conditions.
Time Frame: 48 months
Population: one child did not complete this test. Average age that the children reached a ceiling effect occurred at 30 months (SE: 3.19)
Measure: Mean (Standard Error); unit: percentage of words correct
Arm/Group | Hybrid L24 and Standard CI
Number analyzed (Participants) | 8
percentage of words correct
  Left Ear | 98 (.73)
  Right Ear | 98 (1.71)
  Bilateral | 97 (2.11)

3. Primary Outcome: Phonetically Balanced-Kindergarten
Description: The PB-K test has multiple 50-word lists. The test will be scored as total number of words correct as well as phonemically. It will be administered in both the unilateral and bilateral listening conditions at 70 dB C. Test is administered age-appropriately through study completion.
Time Frame: 60 months
Population: one child withdrew before testing was completed. Average age of testing was 61 mos. (SE: 2.65)
Measure: Mean (Standard Error); unit: percentage of words correct
Arm/Group | Hybrid L24 and Standard CI
Number analyzed (Participants) | 8
percentage of words correct
  Right Ear: number analyzed (Participants) | 7
  Right Ear | 80 (3.5)
  Left Ear | 78 (4.5)
  Bilateral: number analyzed (Participants) | 5
  Bilateral | 81 (5.6)

ADVERSE EVENTS:
Time Frame: activation, 2 weeks, 1 mo., 3 mos., 6 mos., 12 mos., 24 mos., 36 mos., 48 mos., 60 mos.
Arm/Group | Hybrid L24 and Standard CI
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT03156465/Prot_SAP_000.pdf